CLINICAL TRIAL: NCT06416215
Title: Promoting Positive Mental Health for Sustainable Eating Behaviors: the PROMISE Study in Patients With Obesity
Brief Title: Promoting Positive Mental Health for Sustainable Eating Behaviors
Acronym: PROMISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bologna (Other)
Collaborators: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other); European Union (Other)
Responsible Party: Principal Investigator, Elena Tomba, Associate Professor, University of Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROMISE_BO_2024
Record Dates: First submitted 2024-05-09; First posted 2024-05-16 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Cognitive Restructuring

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychological intervention based on WBT and cognitive restructuring (Experimental): Six weekly online sessions of two hours of a psychological intervention based on WBT elements and cognitive restructuring combined with a nutritional education.
  Interventions: Other: Psychological intervention based on WBT and cognitive restructuring
- Basic Nutritional Intervention (Active Comparator): Six weekly online sessions of two hours of a nutritional education.
  Interventions: Other: Basic Nutritional Intervention

INTERVENTIONS:
Other: Psychological intervention based on WBT and cognitive restructuring — Participants will engage in 6 weekly group session of two hours. One part will be held by a trained dietician and will focus on nutritional education, particularly emphasizing the adoption of healthy and sustainable eating behaviors. The remaining part will be dedicated to a group psychological intervention inspired by the principles of Well-Being Therapy and will be held by a trained psychologist. During these sessions, participants will be introduced to the six dimensions of psychological well-being and will be gradually provided with cognitive-behavioral strategies to enhance psychological well-being and seek a balance between the presented dimensions. Participants will be given cognitive-behavioral tools to recognize justification cognitive mechanisms and replace them with more functional cognitions. These objectives will also be achieved through the use of a food diary to highlight emotions and thoughts experienced during food intake.
  Arms: Psychological intervention based on WBT and cognitive restructuring
Other: Basic Nutritional Intervention — Participants will receive treatment as usual (TAU) by participating in 6 weekly group sessions of two hours of a Basic Nutritional Intervention (BNI) held by a trained dietician. This course focuses on promoting healthier lifestyles through nutritional education, diet monitoring using a dedicated food diary, and recommendations for proper physical activity.
  Arms: Basic Nutritional Intervention

SUMMARY:
The main aim of the present study is to assess the effects and the effectiveness of a psychological intervention based on the principles of well-being therapy (WBT) in promoting weight-loss, sustainable and healthy eating behaviors and an optimal psychological functioning in patients with obesity.

DETAILED DESCRIPTION:
The primary objective of this pilot study is to assess the effects and the effectiveness, both post-treatment and at 1- and 3-month follow-ups, of a group intervention inspired by the principles of Well-Being Therapy (WBT), combined with a nutritional education, compared to treatment as usual (TAU), namely a Basic Nutritional Intervention (BNI) in a group setting, in terms of weight loss.

The secondary objective is to evaluate the effects and effectiveness of this intervention, both post-treatment and at 1- and 3-month follow-ups, compared to BNI, in promoting healthy and sustainable eating behaviors and an optimal psychological functioning. This includes the promotion of balanced psychological well-being levels and functional eating styles, and the reduction of both psychological distress and dysfunctional justification cognitive mechanisms use.

After being informed about the study and its potential risks, all patients giving written informed consent will be randomly assigned to either the experimental group or the control group. Both groups will participate in five weekly online group sessions of two hours each.

ELIGIBILITY:
INCLUSION CRITERIA

Patients are included in the study if they:

1. are affiliated with the Clinical Nutrition and Metabolism Unit of Policlinico S. Orsola-Malpighi;
2. have a BMI ≥ 30;
3. are aged ≥ 18 years;
4. voluntarily agree to participate in the study;
5. have access to a computer and can use it independently.

EXCLUSION CRITERIA

Patients are excluded from the study if they:

1. do not sign the informed consent to participate in the study;
2. have limited knowledge of the Italian language;
3. have cognitive deficits;
4. meet the diagnostic criteria for one or more of the following psychiatric diagnoses: drug and/or alcohol abuse, psychotic disorders, neuro-cognitive disorders, suicidal behaviors;
5. participate in another weight loss study or program;
6. take weight loss medications;
7. engage in individual or group psychotherapeutic interventions;
8. have undergone weight loss surgery in the 16 months preceding the study and during the entire study period (approximately five months);
9. (only women) were/are pregnant or were/are planning pregnancy in the 16 months preceding the study and during the entire study period (approximately five months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in weight-loss | Baseline, 35 days after starting the intervention, 1 month after finishing the intervention and 3 months after finishing the intervention
  Body weight will be both self-evaluated by patients and will be verified by the medical staff during follow-up visits

SECONDARY OUTCOMES:
Change from baseline in the Sustainable and Healthy Dietary Behaviors (SHDB) questionnaire | Baseline, 35 days after starting the intervention, 1 month after finishing the intervention and 3 months after finishing the intervention
  The Sustainable and Healthy Dietary Behaviors (SHDB) is 30-item self-reported questionnaire on a 6-point Likert scale to assess sustainable and healthy dietary behaviors through five dimensions and the total score: food choices, storing, cooking, food consumption and food disposal. For each sub-scale and the total score, scores range from 0 to 6, with higher scores indicating more sustainable and healthy eating behaviors (better outcome).
Change from baseline in the Psychological Well-Being Scale (PWBs) | Baseline, 35 days after starting the intervention, 1 month after finishing the intervention and 3 months after finishing the intervention
  The Psychological Well-Being Scale (PWBs) is a 42-item self-reported questionnaire on a 6-point Likert scale that assesses psychological well-being through six dimensions: autonomy, personal growth, environmental mastery, purpose in life, acceptance and positive relations with others. For each dimension scores range from 14 to 84, with higher scores indicating higher levels on that specific PWB dimension (better outcome).
Change from baseline in the Dutch Eating Behavior Questionnaire (DEBQ) | Baseline, 35 days after starting the intervention, 1 month after finishing the intervention and 3 months after finishing the intervention
  The Dutch Eating Behavior Questionnaire (DEBQ) is 33-item self-reported questionnaire on a 5-point Likert scale to assess eating styles through three sub-scales: restrictive eating, emotional eating and external eating.
  For each sub-scale scores range from 1 to 5, with higher scores indicating higher levels on that specific dimension (worse outcome).
Change from baseline in the Depression and Anxiety Stress Scale (DASS-21) | Baseline, 35 days after starting the intervention, 1 month after finishing the intervention and 3 months after finishing the intervention
  The Depression and Anxiety Stress Scale (DASS-21) is a 21-item self-reported questionnaire on a 4-point Likert scale to assess psychological distress through three subscales: depression, anxiety and stress.
  For each sub-scale scores range from 0 to 56, with higher scores indicating higher levels on that specific dimension (worse outcome).
Change from baseline in the use of dysfunctional cognitive justification mechanisms assessed through an ad-hoc form | Baseline, 35 days after starting the intervention, 1 month after finishing the intervention and 3 months after finishing the intervention
  An ad-hoc assessment index adapted from a previous study will be used to assess dysfunctional cognitive justification mechanisms through the presentation of three hypothetical scenarios that could pose dilemmas regarding the adherence to a healthy diet. Participants will be asked to assess their level of identification with the scenario (from 1 to 10) and to specify the type of justification most frequently used in similar situations.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Tomba, Study Director — University of Bologna; Maria Letizia Petroni, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS-S. Orsola-Malpighi Hospital, University of Bologna,, Bologna, Italy

REFERENCES:
- [Result] GBD 2015 Obesity Collaborators; Afshin A, Forouzanfar MH, Reitsma MB, Sur P, Estep K, Lee A, Marczak L, Mokdad AH, Moradi-Lakeh M, Naghavi M, Salama JS, Vos T, Abate KH, Abbafati C, Ahmed MB, Al-Aly Z, Alkerwi A, Al-Raddadi R, Amare AT, Amberbir A, Amegah AK, Amini E, Amrock SM, Anjana RM, Arnlov J, Asayesh H, Banerjee A, Barac A, Baye E, Bennett DA, Beyene AS, Biadgilign S, Biryukov S, Bjertness E, Boneya DJ, Campos-Nonato I, Carrero JJ, Cecilio P, Cercy K, Ciobanu LG, Cornaby L, Damtew SA, Dandona L, Dandona R, Dharmaratne SD, Duncan BB, Eshrati B, Esteghamati A, Feigin VL, Fernandes JC, Furst T, Gebrehiwot TT, Gold A, Gona PN, Goto A, Habtewold TD, Hadush KT, Hafezi-Nejad N, Hay SI, Horino M, Islami F, Kamal R, Kasaeian A, Katikireddi SV, Kengne AP, Kesavachandran CN, Khader YS, Khang YH, Khubchandani J, Kim D, Kim YJ, Kinfu Y, Kosen S, Ku T, Defo BK, Kumar GA, Larson HJ, Leinsalu M, Liang X, Lim SS, Liu P, Lopez AD, Lozano R, Majeed A, Malekzadeh R, Malta DC, Mazidi M, McAlinden C, McGarvey ST, Mengistu DT, Mensah GA, Mensink GBM, Mezgebe HB, Mirrakhimov EM, Mueller UO, Noubiap JJ, Obermeyer CM, Ogbo FA, Owolabi MO, Patton GC, Pourmalek F, Qorbani M, Rafay A, Rai RK, Ranabhat CL, Reinig N, Safiri S, Salomon JA, Sanabria JR, Santos IS, Sartorius B, Sawhney M, Schmidhuber J, Schutte AE, Schmidt MI, Sepanlou SG, Shamsizadeh M, Sheikhbahaei S, Shin MJ, Shiri R, Shiue I, Roba HS, Silva DAS, Silverberg JI, Singh JA, Stranges S, Swaminathan S, Tabares-Seisdedos R, Tadese F, Tedla BA, Tegegne BS, Terkawi AS, Thakur JS, Tonelli M, Topor-Madry R, Tyrovolas S, Ukwaja KN, Uthman OA, Vaezghasemi M, Vasankari T, Vlassov VV, Vollset SE, Weiderpass E, Werdecker A, Wesana J, Westerman R, Yano Y, Yonemoto N, Yonga G, Zaidi Z, Zenebe ZM, Zipkin B, Murray CJL. Health Effects of Overweight and Obesity in 195 Countries over 25 Years. N Engl J Med. 2017 Jul 6;377(1):13-27. doi: 10.1056/NEJMoa1614362. Epub 2017 Jun 12. PMID 28604169
- [Result] Aguera Z, Lozano-Madrid M, Mallorqui-Bague N, Jimenez-Murcia S, Menchon JM, Fernandez-Aranda F. A review of binge eating disorder and obesity. Neuropsychiatr. 2021 Jun;35(2):57-67. doi: 10.1007/s40211-020-00346-w. Epub 2020 Apr 28. PMID 32346850
- [Result] Alimoradi Z, Golboni F, Griffiths MD, Brostrom A, Lin CY, Pakpour AH. Weight-related stigma and psychological distress: A systematic review and meta-analysis. Clin Nutr. 2020 Jul;39(7):2001-2013. doi: 10.1016/j.clnu.2019.10.016. Epub 2019 Oct 31. PMID 31732288
- [Result] Bischoff SC, Boirie Y, Cederholm T, Chourdakis M, Cuerda C, Delzenne NM, Deutz NE, Fouque D, Genton L, Gil C, Koletzko B, Leon-Sanz M, Shamir R, Singer J, Singer P, Stroebele-Benschop N, Thorell A, Weimann A, Barazzoni R. Towards a multidisciplinary approach to understand and manage obesity and related diseases. Clin Nutr. 2017 Aug;36(4):917-938. doi: 10.1016/j.clnu.2016.11.007. Epub 2016 Nov 16. PMID 27890486
- [Result] Bottesi G, Ghisi M, Altoe G, Conforti E, Melli G, Sica C. The Italian version of the Depression Anxiety Stress Scales-21: Factor structure and psychometric properties on community and clinical samples. Compr Psychiatry. 2015 Jul;60:170-81. doi: 10.1016/j.comppsych.2015.04.005. Epub 2015 Apr 15. PMID 25933937
- [Result] Brantley PJ, Stewart DW, Myers VH, Matthews-Ewald MR, Ard JD, Coughlin JW, Jerome GJ, Samuel-Hodge C, Lien LF, Gullion CM, Hollis JF, Svetkey LP, Stevens VJ. Psychosocial predictors of weight regain in the weight loss maintenance trial. J Behav Med. 2014 Dec;37(6):1155-68. doi: 10.1007/s10865-014-9565-6. Epub 2014 Apr 11. PMID 24722826
- [Result] Castelnuovo G, Pietrabissa G, Manzoni GM, Corti S, Ceccarini M, Borrello M, Giusti EM, Novelli M, Cattivelli R, Middleton NA, Simpson SG, Molinari E. Chronic care management of globesity: promoting healthier lifestyles in traditional and mHealth based settings. Front Psychol. 2015 Oct 15;6:1557. doi: 10.3389/fpsyg.2015.01557. eCollection 2015. PMID 26528215
- [Result] Chu DT, Minh Nguyet NT, Dinh TC, Thai Lien NV, Nguyen KH, Nhu Ngoc VT, Tao Y, Son LH, Le DH, Nga VB, Jurgonski A, Tran QH, Van Tu P, Pham VH. An update on physical health and economic consequences of overweight and obesity. Diabetes Metab Syndr. 2018 Nov;12(6):1095-1100. doi: 10.1016/j.dsx.2018.05.004. Epub 2018 May 5. PMID 29799416
- [Result] da Luz FQ, Hay P, Touyz S, Sainsbury A. Obesity with Comorbid Eating Disorders: Associated Health Risks and Treatment Approaches. Nutrients. 2018 Jun 27;10(7):829. doi: 10.3390/nu10070829. PMID 29954056
- [Result] Dakanalis A, Zanetti MA, Clerici M, Madeddu F, Riva G, Caccialanza R. Italian version of the Dutch Eating Behavior Questionnaire. Psychometric proprieties and measurement invariance across sex, BMI-status and age. Appetite. 2013 Dec;71:187-95. doi: 10.1016/j.appet.2013.08.010. Epub 2013 Aug 30. PMID 23994503
- [Result] Fava GA. Well-being therapy: Treatment manual and clinical applications. Karger Medical and Scientific Publishers. 2016
- [Result] Fava GA. Well-Being Therapy: Current Indications and Emerging Perspectives. Psychother Psychosom. 2016;85(3):136-45. doi: 10.1159/000444114. Epub 2016 Apr 5. No abstract available. PMID 27043240
- [Result] Fischer M, Oberander N, Weimann A. Four main barriers to weight loss maintenance? A quantitative analysis of difficulties experienced by obese patients after successful weight reduction. Eur J Clin Nutr. 2020 Aug;74(8):1192-1200. doi: 10.1038/s41430-020-0559-x. Epub 2020 Jan 30. PMID 32001814
- [Result] Hudson JI, Hiripi E, Pope HG Jr, Kessler RC. The prevalence and correlates of eating disorders in the National Comorbidity Survey Replication. Biol Psychiatry. 2007 Feb 1;61(3):348-58. doi: 10.1016/j.biopsych.2006.03.040. Epub 2006 Jul 3. PMID 16815322
- [Result] Kantartzis K, Machann J, Schick F, Rittig K, Machicao F, Fritsche A, Haring HU, Stefan N. Effects of a lifestyle intervention in metabolically benign and malign obesity. Diabetologia. 2011 Apr;54(4):864-8. doi: 10.1007/s00125-010-2006-3. Epub 2010 Dec 21. PMID 21174075
- [Result] Kawasaki Y, Nagao-Sato S, Yoshii E, Akamatsu R. Integrated consumers' sustainable and healthy dietary behavior patterns: Associations between demographics, psychological factors, and meal preparation habits among Japanese adults. Appetite. 2023 Jan 1;180:106353. doi: 10.1016/j.appet.2022.106353. Epub 2022 Oct 26. PMID 36309231
- [Result] Lillis J, Kendra KE. Acceptance and Commitment Therapy for weight control: Model, evidence, and future directions. J Contextual Behav Sci. 2014 Jan;3(1):1-7. doi: 10.1016/j.jcbs.2013.11.005. PMID 25419510
- [Result] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Result] Mantzios M, Egan HH. On the Role of Self-compassion and Self-kindness in Weight Regulation and Health Behavior Change. Front Psychol. 2017 Feb 16;8:229. doi: 10.3389/fpsyg.2017.00229. eCollection 2017. No abstract available. PMID 28261147
- [Result] Manzoni GM, Cribbie RA, Villa V, Arpin-Cribbie CA, Gondoni L, Castelnuovo G. Psychological well-being in obese inpatients with ischemic heart disease at entry and at discharge from a four-week cardiac rehabilitation program. Front Psychol. 2010 Aug 3;1:38. doi: 10.3389/fpsyg.2010.00038. eCollection 2010. PMID 21833207
- [Result] Popkin BM, Ng SW. The nutrition transition to a stage of high obesity and noncommunicable disease prevalence dominated by ultra-processed foods is not inevitable. Obes Rev. 2022 Jan;23(1):e13366. doi: 10.1111/obr.13366. Epub 2021 Oct 10. PMID 34632692
- [Result] Ruini C, Ottolini F, Rafanelli C, Ryff CD, Fava GA. La validazione italiana delle Psychological Well-being Scales (PWB). Rivista di psichiatria. 2003; 38(3): 117-130.
- [Result] Ryff CD, Singer B. Psychological well-being: meaning, measurement, and implications for psychotherapy research. Psychother Psychosom. 1996;65(1):14-23. doi: 10.1159/000289026. PMID 8838692
- [Result] Sarwer DB, Allison KC, Wadden TA, Ashare R, Spitzer JC, McCuen-Wurst C, LaGrotte C, Williams NN, Edwards M, Tewksbury C, Wu J. Psychopathology, disordered eating, and impulsivity as predictors of outcomes of bariatric surgery. Surg Obes Relat Dis. 2019 Apr;15(4):650-655. doi: 10.1016/j.soard.2019.01.029. Epub 2019 Feb 23. PMID 30858009
- [Result] Sharma M. Behavioural interventions for preventing and treating obesity in adults. Obes Rev. 2007 Sep;8(5):441-9. doi: 10.1111/j.1467-789X.2007.00351.x. PMID 17716301
- [Result] Taylor C, Webb TL, Sheeran P. 'I deserve a treat!': justifications for indulgence undermine the translation of intentions into action. Br J Soc Psychol. 2014 Sep;53(3):501-20. doi: 10.1111/bjso.12043. Epub 2013 Jul 15. PMID 23855962
- [Result] Teixeira PJ, Going SB, Houtkooper LB, Cussler EC, Metcalfe LL, Blew RM, Sardinha LB, Lohman TG. Pretreatment predictors of attrition and successful weight management in women. Int J Obes Relat Metab Disord. 2004 Sep;28(9):1124-33. doi: 10.1038/sj.ijo.0802727. PMID 15263921
- [Result] Turton R, Chami R, Treasure J. Emotional Eating, Binge Eating and Animal Models of Binge-Type Eating Disorders. Curr Obes Rep. 2017 Jun;6(2):217-228. doi: 10.1007/s13679-017-0265-8. PMID 28434108
- [Result] Van Strien T, Frijters JE, Bergers GP, Defares PB. The Dutch Eating Behavior Questionnaire (DEBQ) for assessment of restrained, emotional, and external eating behavior. International journal of eating disorders. 1986; 5(2): 295-315.
- [Result] Vallis M. Quality of life and psychological well-being in obesity management: improving the odds of success by managing distress. Int J Clin Pract. 2016 Mar;70(3):196-205. doi: 10.1111/ijcp.12765. Epub 2016 Feb 4. PMID 26842304
- [Result] Webber KH, Casey EM, Mayes L, Katsumata Y, Mellin L. A comparison of a behavioral weight loss program to a stress management program: A pilot randomized controlled trial. Nutrition. 2016 Jul-Aug;32(7-8):904-9. doi: 10.1016/j.nut.2016.01.008. Epub 2016 Jan 21. PMID 27138110
- [Result] Zhu B, Gostoli S, Benasi G, Patierno C, Petroni ML, Nuccitelli C, Marchesini G, Fava GA, Rafanelli C. Promoting weight loss and psychological well-being in patients with obesity: A sequential combination of behavioural lifestyle intervention and well-being therapy. Clin Psychol Psychother. 2023 Mar;30(2):422-435. doi: 10.1002/cpp.2806. Epub 2022 Dec 20. PMID 36436883

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-21): https://cdn.clinicaltrials.gov/large-docs/15/NCT06416215/Prot_SAP_000.pdf